CLINICAL TRIAL: NCT00738894
Title: GORE® HELEX® Septal Occluder / GORE® CARDIOFORM Septal Occluder and Antiplatelet Medical Management for Reduction of Recurrent Stroke or Imaging-Confirmed TIA in Patients With Patent Foramen Ovale (PFO) - The Gore REDUCE Clinical Study
Brief Title: GORE® Septal Occluder Device for Patent Foramen Ovale (PFO) Closure in Stroke Patients
Acronym: REDUCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HLX 06-03
Record Dates: First submitted 2008-08-19; First posted 2008-08-21 (Estimated); Results first posted 2018-08-09 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-10

CONDITIONS: Stroke; Transient Ischemic Attack
Keywords: cryptogenic; stroke; transient ischemic attack; TIA; PFO; Patent foramen ovale; HELEX; Septal Occluder; PFO Occluder
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Foramen Ovale, Patent | interventions — Septal Occluder Device; Aspirin; Dipyridamole; Aspirin, Dipyridamole Drug Combination; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medical Management (Active Comparator): Antiplatelet medical therapy alone
  Interventions: Drug: Antiplatelet Medical Therapy
- Device Closure (Experimental): PFO closure with study septal occluder device plus antiplatelet medical therapy
  Interventions: Device: Septal Occluder Device; Drug: Antiplatelet Medical Therapy

INTERVENTIONS:
Device: Septal Occluder Device — PFO closure with study septal occluder device
  Other Names: GORE® HELEX® Septal Occluder; GORE® CARDIOFORM Septal Occluder
  Arms: Device Closure
Drug: Antiplatelet Medical Therapy — Investigator's choice of one of three regimen options specified in protocol
  Other Names: Aspirin; Dipyridamole; Aggrenox; Clopidogrel; Plavix

SUMMARY:
The primary objective is to determine if patent foramen ovale (PFO) closure with the GORE® HELEX® Septal Occluder or GORE® CARDIOFORM Septal Occluder plus antiplatelet medical management is safe and effective and reduces the risk of recurrent stroke or imaging-confirmed transient ischemic attack (TIA) when compared to antiplatelet medical management alone in patients with a PFO and history of cryptogenic stroke or imaging-confirmed TIA.

A co-primary objective is to demonstrate that medical management plus closure with the study device reduces the risk of new brain infarct compared to medical management alone.

ELIGIBILITY:
Inclusion Criteria:

* Presence of cryptogenic ischemic stroke or TIA of presumed embolic infarction verified by a neurologist within 180 days prior to randomization
* Presence of Patent Foramen Ovale (PFO), as determined initially by positive bubble study utilizing transesophageal echocardiography (TEE), demonstrating spontaneous right-to-left shunting or right-to-left shunting during Valsalva maneuver.
* Absence of an identifiable source of thromboembolism in the systemic circulation
* No evidence of a hypercoagulable state
* Note: Additional Inclusion Criteria may apply

Exclusion Criteria:

* Other co-morbidities including, but not limited to, mural thrombus, dilated cardiomyopathy, atrial fibrillation/flutter, cardiac prosthetics (valves), mitral valve stenosis, aortic dissection, significant atherosclerosis, vasculitis, pre-existing neurologic disorders, multiple sclerosis, arteriovenous malformations, prior intracranial hemorrhage, severe central nervous system (CNS) disease, severe disability related to prior stroke, and autoimmune disorders that would increase the risk of mortality or morbidity above what is typical for the treatment
* Previous Myocardial Infarction
* Active infection that cannot be treated successfully prior to randomization
* Sensitivity or contraindication to all proposed medical treatments
* Pregnancy or intent on becoming pregnant through 24-months after randomization
* Indications outside the parameters accepted for placement of the GORE® HELEX® Septal Occluder / GORE® Septal Occluder, including extensive congenital cardiac anomalies and defect diameter estimated to be > 18mm
* Atrial septal anatomy that is expected to necessitate placement of more than one GORE® HELEX® Septal Occluder / GORE® CARDIOFORM Septal Occluder
* Need for concomitant procedure(s) that may confound detection of adverse events related to device placement
* Note: Additional Exclusion Criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 664 (Actual)
Dates: Start 2008-12-10 (Actual); Primary Completion 2017-04-24 (Actual); Study Completion 2020-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott E. Kasner, MD, FAHA, Principal Investigator — University of Pennsylvania Medical Center; John F. Rhodes, MD, Principal Investigator — Medical University of South Carolina; Lars Søndergaard, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- University of Pennsylvania Medical Center, Philadelphia, Pennsylvania, United States
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Messe SR, Erus G, Bilello M, Davatzikos C, Andersen G, Iversen HK, Roine RO, Sjostrand C, Rhodes JF, Sondergaard L, Kasner SE; Gore REDUCE Study Investigators. Patent Foramen Ovale Closure Decreases the Incidence but Not the Size of New Brain Infarction on Magnetic Resonance Imaging: An Analysis of the REDUCE Trial. Stroke. 2021 Nov;52(11):3419-3426. doi: 10.1161/STROKEAHA.121.034451. Epub 2021 Aug 30. PMID 34455822
- [Derived] Kasner SE, Thomassen L, Sondergaard L, Rhodes JF, Larsen CC, Jacobson J. Patent foramen ovale closure with GORE HELEX or CARDIOFORM Septal Occluder vs. antiplatelet therapy for reduction of recurrent stroke or new brain infarct in patients with prior cryptogenic stroke: Design of the randomized Gore REDUCE Clinical Study. Int J Stroke. 2017 Dec;12(9):998-1004. doi: 10.1177/1747493017701152. Epub 2017 Mar 24. PMID 29090661
- [Derived] Sondergaard L, Kasner SE, Rhodes JF, Andersen G, Iversen HK, Nielsen-Kudsk JE, Settergren M, Sjostrand C, Roine RO, Hildick-Smith D, Spence JD, Thomassen L; Gore REDUCE Clinical Study Investigators. Patent Foramen Ovale Closure or Antiplatelet Therapy for Cryptogenic Stroke. N Engl J Med. 2017 Sep 14;377(11):1033-1042. doi: 10.1056/NEJMoa1707404. PMID 28902580

RESULTS

PARTICIPANT FLOW:
Groups:
- Device Closure: PFO closure with study septal occluder device plus antiplatelet medical therapy
  Septal Occluder Device: GORE® HELEX® Septal Occluder or GORE® CARDIOFORM Septal Occluder
  Antiplatelet Medical Therapy: Investigator's choice of one of three regimen options specified in protocol
Period: Overall Study
Arm/Group | Device Closure | Medical Management
Started | 441 | 223
Completed | 402 | 190
Not Completed | 39 | 33
Not completed — Lost to Follow-up | 23 | 13
Not completed — Withdrawal by Subject | 10 | 15
Not completed — Physician Decision | 4 | 5
Not completed — Death | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Device Closure | Medical Management | Total
Number analyzed (Participants) | 441 | 223 | 664
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (9.3) | 44.8 (9.6) | 45.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180 | 85 | 265
  Male | 261 | 138 | 399
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 9 | 31
  Not Hispanic or Latino | 413 | 213 | 626
  Unknown or Not Reported | 6 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 12 | 26
  White | 412 | 203 | 615
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 10 | 5 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 216 | 115 | 331
  Canada | 17 | 8 | 25
  Denmark | 79 | 38 | 117
  Finland | 18 | 8 | 26
  Norway | 25 | 14 | 39
  Sweden | 64 | 31 | 95
  United Kingdom | 22 | 9 | 31
Time from qualifying event to randomization [Mean (Standard Deviation); unit: days] | 100 (52) | 101 (53) | 101 (53)
Current smoking [Count of Participants; unit: Participants] | 63 | 25 | 88
Hypertension [Count of Participants; unit: Participants] | 112 | 58 | 170
Diabetes mellitus [Count of Participants; unit: Participants] | 18 | 10 | 28
Stroke or TIA before index event [Count of Participants; unit: Participants]
  Previous either | 62 | 23 | 85
  Previous stroke | 42 | 13 | 55
  Previous TIA | 26 | 11 | 37
Index event [Count of Participants; unit: Participants]
  Stroke w/ symptoms >=24 hr | 402 | 199 | 601
  Stroke symptoms <24 hr, w/ imaging confirmation | 39 | 24 | 63
Patent foramen ovale shunt size [Count of Participants; unit: Participants] — Population: 16 device closure subjects and 7 medical management subjects reported shunt assessment of unknown, unable to perform, or not performed.
  Participants
    number analyzed (Participants) | 425 | 216 | 641
    Small (1-5 bubbles) | 77 | 43 | 120
    Moderate (6-25 bubbles) | 166 | 94 | 260
    Large (>25 bubbles) | 182 | 79 | 261
Atrial septal aneurysm [Count of Participants; unit: Participants] — Population: Atrial septal aneurysm was determined during the PFO closure procedure; it was not recorded for any medical management subjects, nor for 19 of the 28 device closure subjects with no study device implant attempt.
  Participants
    number analyzed (Participants) | 422 | 0 | 422
    (all) | 86 |  | 86

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Freedom From Recurrent Ischemic Stroke (Primary Outcome #1)
Description: A recurrent stroke event was defined as the first occurrence post-randomization of either a) neurological deficit presumed due to ischemia and persisting longer than 24 hours or until death, or b) transient neurological deficit presumed due to ischemia, persisting less than 24 hours with MRI evidence of a new relevant brain infarction.
Time Frame: 24 months
Population: Intention to Treat: includes all subjects randomized
Measure: Count of Participants; unit: Participants
Arm/Group | Device Closure | Medical Management
Number analyzed (Participants) | 441 | 223
Participants | 6 | 12
Statistical Analysis 1: Comparison: Device Closure vs Medical Management; Test null hypothesis of equal or lower recurrent stroke-free survivorship for device closure compared to medical management. H0: Sd(t) ≤ Sm(t) for all t, versus H1: Sd(t) > Sm(t) for all t, where Sd(t) and Sm(t) are true Kaplan-Meier product-limit survivor functions for the device closure and medical management arms and t is time from randomization to event or censoring. Event-free subjects were censored at time of last follow-up. Significance threshold (1-sided alpha) = 0.025; Test type: Superiority — This is the first of two primary outcomes for this study. Assumptions for power calculations: expected event free for medical management 92% at 24 months; expected event free for device closure 96.4% at 24 months (55% risk reduction); 664 subjects randomly assigned 2:1 to device closure or medical management provides 80% power with 15% attrition (over 5 years) and 1-sided alpha = 0.024 to allow for interim analysis (interim analysis later rescinded from plan); p = 0.001, Log Rank — 1-sided p-value was adjusted for multiplicity with 2nd primary outcome using Dubey and Armitage-Parmer (D/AP) procedure; Hazard Ratio (HR) = 0.23, 95% CI 2-sided [0.09 to 0.62] — Hazard ratio (test/control) obtained from Cox proportional hazards model with treatment arm as sole explanatory variable, the exponentiated coefficient of which provided the hazard ratio. Unadjusted for multiplicity

2. Primary Outcome: Number of Subjects With New Brain Infarct or Recurrent Stroke (Primary Outcome #2)
Description: Responders were subjects who showed one or more new infarctions on MRI since screening, or experienced a confirmed recurrent stroke, through 24 months (913 days). Nonresponders were subjects who did not show new infarction on MRI since screening and were confirmed free of recurrent stroke through at least 549 days.
  An infarction was defined as a new (since screening) T2 hyperintense MRI lesion with diameter ≥ 3 mm.
Time Frame: 24 months
Population: Intention to Treat: includes all subjects randomized and evaluated for brain infarct
Measure: Count of Participants; unit: Participants
Arm/Group | Device Closure | Medical Management
Number analyzed (Participants) | 383 | 177
Participants | 22 | 20
Statistical Analysis 1: Comparison: Device Closure vs Medical Management; Test null hypothesis of equal or higher proportion with brain infarct for device closure compared to medical management. H0: Pm - Pd ≤ 0, versus H1: Pm - Pd > 0, where Pd and Pm are true proportions of subjects with brain infarct for the device closure and medical management arms. Significance threshold (1-sided alpha) = 0.025; Test type: Superiority — This is the second of two primary outcomes for this study. Assumptions for power calculations: expected proportion of brain infarct is 3-7 times the clinical stroke rate; expected brain infarct proportion for medical management 14.5% (2.9% clinical stroke x 5); expected brain infarct for device closure 6.5% (55% risk reduction); 597 subjects (10% attrition from 664) provides 73% power with 1-sided alpha = 0.0125 (based conservatively on a Bonferroni adjustment of alpha/2); p = 0.024, z-test, 1-sided — 1-sided p-value was adjusted for multiplicity with 1st primary outcome using Dubey and Armitage-Parmer (D/AP) procedure; Risk Difference (RD) = 0.056, 95% CI 2-sided [0.003 to 0.108] — Unadjusted for multiplicity

3. Secondary Outcome: Number of Subjects With Study-related Serious Adverse Events
Description: Adverse event seriousness and relationship to study treatments (device, procedure, or antiplatelet medical therapy) as reported by each investigative site
Time Frame: 24 months
Population: Intention to Treat: all subjects randomized
Measure: Count of Participants; unit: Participants
Arm/Group | Device Closure | Medical Management
Number analyzed (Participants) | 441 | 223
Participants | 102 | 62

4. Secondary Outcome: Number of Subjects With Effective Closure in Test (Device) Arm
Description: Assessment of PFO closure in test (device) arm subjects by transesophageal echocardiography (TEE) at 24-month follow-up.
  Effective closure defined as occluded, small, or moderate shunt (0-25 bubbles).
Time Frame: 24 months
Population: All subjects randomized to test (device) arm with 24-month PFO closure assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Device Closure
Number analyzed (Participants) | 318
Participants | 312

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Device Closure | Medical Management
All-Cause Mortality (participants affected / at risk) | 2/441 | 0/223
Serious Adverse Events (participants affected / at risk) | 102/441 | 62/223
Other Adverse Events (participants affected / at risk) | 324/441 | 154/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Device Closure (N=441) | Medical Management (N=223)
Headache (Nervous system disorders) | 6 | 4
Cerebrovascular accident (Nervous system disorders) | 4 | 5
Transient ischaemic attack (Nervous system disorders) | 4 | 5
Dizziness (Nervous system disorders) | 4 | 4
Dysaesthesia (Nervous system disorders) | 6 | 2
Migraine with aura (Nervous system disorders) | 5 | 3
Syncope (Nervous system disorders) | 2 | 4
Paraesthesia (Nervous system disorders) | 2 | 2
Migraine (Nervous system disorders) | 2 | 1
Carotid artery dissection (Nervous system disorders) | 1 | 1
Cerebral infarction (Nervous system disorders) | 1 | 1
Dysarthria (Nervous system disorders) | 1 | 1
Hemiparesis (Nervous system disorders) | 2 | 0
Monoparesis (Nervous system disorders) | 1 | 1
Aphasia (Nervous system disorders) | 1 | 0
Diabetic hyperosmolar coma (Nervous system disorders) | 0 | 1
Dural arteriovenous fistula (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Lacunar infarction (Nervous system disorders) | 0 | 1
Nystagmus (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Tension headache (Nervous system disorders) | 0 | 1
Thunderclap headache (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Ulnar tunnel syndrome (Nervous system disorders) | 0 | 1
Vertebral artery dissection (Nervous system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 10 | 1
Palpitations (Cardiac disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Pericardial cyst (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Pulseless electrical activity (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 2
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Incision site complication (Injury, poisoning and procedural complications) | 1 | 0
Incision site haematoma (Injury, poisoning and procedural complications) | 1 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Appendicitis (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 1 | 2
Campylobacter infection (Infections and infestations) | 1 | 0
Chronic tonsillitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Malaria (Infections and infestations) | 1 | 0
Renal abscess (Infections and infestations) | 0 | 1
Staphylococcal skin infection (Infections and infestations) | 1 | 0
Streptococcal infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Viral pericarditis (Infections and infestations) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 2 | 0
Aortic dissection (Vascular disorders) | 1 | 0
Arteriovenous fistula (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral embolism (Vascular disorders) | 0 | 1
Vena cava thrombosis (Vascular disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 3 | 1
Fatigue (General disorders) | 2 | 1
Adverse drug reaction (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Complication of device removal (General disorders) | 1 | 0
Puncture site haemorrhage (General disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 2
Bipolar disorder (Psychiatric disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Conversion disorder (Psychiatric disorders) | 0 | 1
Delusion (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0
Mania (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Paranoia (Psychiatric disorders) | 1 | 0
Schizoaffective disorder (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 2
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Biliary colic (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 4 | 1
Blindness unilateral (Eye disorders) | 0 | 1
Eye haemorrhage (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 1
Device dislocation (Product Issues) | 3 | 0
Thrombosis in device (Product Issues) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 3 | 0
Calculus urethral (Renal and urinary disorders) | 0 | 1
Urethral meatus stenosis (Renal and urinary disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Adrenal mass (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Osteosynthesis (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Device Closure (N=441) | Medical Management (N=223)
Headache (Nervous system disorders) | 37 | 32
Dizziness (Nervous system disorders) | 34 | 16
Dysaesthesia (Nervous system disorders) | 19 | 19
Migraine (Nervous system disorders) | 15 | 5
Migraine with aura (Nervous system disorders) | 8 | 4
Transient ischaemic attack (Nervous system disorders) | 6 | 5
Paraesthesia (Nervous system disorders) | 10 | 3
Cerebrovascular accident (Nervous system disorders) | 1 | 4
Syncope (Nervous system disorders) | 5 | 2
Memory impairment (Nervous system disorders) | 5 | 4
Dysarthria (Nervous system disorders) | 3 | 2
Monoparesis (Nervous system disorders) | 3 | 2
Presyncope (Nervous system disorders) | 7 | 0
Aphasia (Nervous system disorders) | 1 | 4
Hemiparesis (Nervous system disorders) | 3 | 1
Seizure (Nervous system disorders) | 2 | 2
Balance disorder (Nervous system disorders) | 2 | 2
Cervical radiculopathy (Nervous system disorders) | 3 | 1
Facial paralysis (Nervous system disorders) | 2 | 2
Visual field defect (Nervous system disorders) | 2 | 2
Amnesia (Nervous system disorders) | 1 | 2
Ataxia (Nervous system disorders) | 1 | 2
Cerebral infarction (Nervous system disorders) | 1 | 0
Disturbance in attention (Nervous system disorders) | 1 | 2
Hypoaesthesia (Nervous system disorders) | 2 | 1
Lumbar radiculopathy (Nervous system disorders) | 1 | 2
Sensory disturbance (Nervous system disorders) | 2 | 1
Tension headache (Nervous system disorders) | 1 | 1
Carpal tunnel syndrome (Nervous system disorders) | 2 | 0
Lacunar infarction (Nervous system disorders) | 0 | 1
Nerve compression (Nervous system disorders) | 1 | 1
Sciatica (Nervous system disorders) | 0 | 1
Sensory loss (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 1 | 0
Amimia (Nervous system disorders) | 1 | 0
Aura (Nervous system disorders) | 1 | 0
Burning sensation (Nervous system disorders) | 0 | 1
Clumsiness (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 1 | 0
Dizziness postural (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Exertional headache (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 1 | 0
Fine motor skill dysfunction (Nervous system disorders) | 1 | 0
Focal dyscognitive seizures (Nervous system disorders) | 1 | 0
Head discomfort (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Mental impairment (Nervous system disorders) | 0 | 1
Morton's neuralgia (Nervous system disorders) | 1 | 0
Muscle spasticity (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Nystagmus (Nervous system disorders) | 0 | 1
Occipital neuralgia (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 1
Pineal gland cyst (Nervous system disorders) | 1 | 0
Quadrantanopia (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Speech disorder (Nervous system disorders) | 1 | 0
Subdural effusion (Nervous system disorders) | 0 | 1
Ulnar neuritis (Nervous system disorders) | 0 | 1
Upper motor neurone lesion (Nervous system disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 23 | 4
Sinusitis (Infections and infestations) | 13 | 6
Bronchitis (Infections and infestations) | 11 | 3
Urinary tract infection (Infections and infestations) | 12 | 2
Influenza (Infections and infestations) | 11 | 1
Nasopharyngitis (Infections and infestations) | 8 | 4
Pneumonia (Infections and infestations) | 5 | 2
Acute sinusitis (Infections and infestations) | 3 | 2
Pharyngitis (Infections and infestations) | 4 | 1
Herpes zoster (Infections and infestations) | 3 | 1
Skin infection (Infections and infestations) | 1 | 3
Chronic tonsillitis (Infections and infestations) | 2 | 0
Cystitis (Infections and infestations) | 2 | 0
Ear infection (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Onychomycosis (Infections and infestations) | 2 | 1
Otitis media (Infections and infestations) | 3 | 0
Cellulitis (Infections and infestations) | 2 | 0
Diverticulitis (Infections and infestations) | 1 | 1
Epididymitis (Infections and infestations) | 1 | 1
Folliculitis (Infections and infestations) | 1 | 1
Otitis externa (Infections and infestations) | 2 | 0
Otitis media acute (Infections and infestations) | 2 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 1
Pyelonephritis (Infections and infestations) | 2 | 0
Subcutaneous abscess (Infections and infestations) | 2 | 0
Tinea pedis (Infections and infestations) | 2 | 0
Tooth infection (Infections and infestations) | 2 | 0
Vaginal infection (Infections and infestations) | 2 | 0
Viral labyrinthitis (Infections and infestations) | 1 | 1
Abscess limb (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Epstein-Barr virus infection (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Eye infection (Infections and infestations) | 0 | 1
Gastroenteritis salmonella (Infections and infestations) | 0 | 1
Groin infection (Infections and infestations) | 1 | 0
Helicobacter infection (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Hordeolum (Infections and infestations) | 1 | 0
Impetigo (Infections and infestations) | 1 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 1
Labyrinthitis (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Oral viral infection (Infections and infestations) | 1 | 0
Otitis media chronic (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 0 | 1
Perichondritis (Infections and infestations) | 0 | 1
Pilonidal cyst (Infections and infestations) | 1 | 0
Rash pustular (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Tinea cruris (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Palpitations (Cardiac disorders) | 64 | 14
Atrial fibrillation (Cardiac disorders) | 21 | 0
Tachycardia (Cardiac disorders) | 10 | 1
Angina pectoris (Cardiac disorders) | 3 | 1
Sinus tachycardia (Cardiac disorders) | 2 | 1
Supraventricular extrasystoles (Cardiac disorders) | 2 | 1
Ventricular extrasystoles (Cardiac disorders) | 3 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Extrasystoles (Cardiac disorders) | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Atrial thrombosis (Cardiac disorders) | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Cardiac discomfort (Cardiac disorders) | 1 | 0
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 5 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 3 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 2 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 2 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Inguinal mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Jaw disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 1 | 0
Myokymia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 11 | 2
Incision site pain (Injury, poisoning and procedural complications) | 9 | 0
Laceration (Injury, poisoning and procedural complications) | 5 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 6 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 6 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 4 | 2
Incision site haematoma (Injury, poisoning and procedural complications) | 5 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 5 | 0
Foot fracture (Injury, poisoning and procedural complications) | 4 | 0
Incision site complication (Injury, poisoning and procedural complications) | 3 | 0
Limb injury (Injury, poisoning and procedural complications) | 4 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 2
Procedural complication (Injury, poisoning and procedural complications) | 3 | 0
Procedural pain (Injury, poisoning and procedural complications) | 3 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 3 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 2 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 2 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 2 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1
Animal scratch (Injury, poisoning and procedural complications) | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 | 0
Exposure to body fluid (Injury, poisoning and procedural complications) | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1
Persistent corneal epithelial defect (Injury, poisoning and procedural complications) | 1 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 | 0
Procedural headache (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Non-cardiac chest pain (General disorders) | 23 | 11
Fatigue (General disorders) | 13 | 9
Chest discomfort (General disorders) | 11 | 2
Oedema peripheral (General disorders) | 10 | 0
Chest pain (General disorders) | 4 | 2
Peripheral swelling (General disorders) | 3 | 3
Adverse drug reaction (General disorders) | 3 | 0
Pyrexia (General disorders) | 2 | 1
Influenza like illness (General disorders) | 1 | 1
Oedema (General disorders) | 1 | 1
Puncture site haemorrhage (General disorders) | 1 | 0
Drug withdrawal syndrome (General disorders) | 1 | 0
Feeling abnormal (General disorders) | 1 | 0
Feeling hot (General disorders) | 0 | 1
Gait disturbance (General disorders) | 1 | 0
Hernia (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Puncture site pain (General disorders) | 1 | 0
Suprapubic pain (General disorders) | 0 | 1
Temperature intolerance (General disorders) | 0 | 1
Thirst (General disorders) | 0 | 1
Vessel puncture site bruise (General disorders) | 1 | 0
Vessel puncture site haemorrhage (General disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 14 | 7
Abdominal pain upper (Gastrointestinal disorders) | 4 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 2
Constipation (Gastrointestinal disorders) | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 2
Abdominal pain (Gastrointestinal disorders) | 4 | 2
Gastritis (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 1
Haematochezia (Gastrointestinal disorders) | 2 | 2
Inguinal hernia (Gastrointestinal disorders) | 2 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 1
Hiatus hernia (Gastrointestinal disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 0
Large intestine polyp (Gastrointestinal disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal wall cyst (Gastrointestinal disorders) | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Change of bowel habit (Gastrointestinal disorders) | 1 | 0
Colitis microscopic (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 1 | 0
Oesophageal pain (Gastrointestinal disorders) | 1 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 1 | 0
Rectal fissure (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 17 | 4
Depression (Psychiatric disorders) | 8 | 8
Insomnia (Psychiatric disorders) | 8 | 5
Post stroke depression (Psychiatric disorders) | 5 | 2
Affect lability (Psychiatric disorders) | 3 | 1
Confusional state (Psychiatric disorders) | 3 | 1
Panic attack (Psychiatric disorders) | 2 | 2
Sleep disorder (Psychiatric disorders) | 0 | 4
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 2 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Agitated depression (Psychiatric disorders) | 1 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Anxiety disorder (Psychiatric disorders) | 1 | 0
Drug abuse (Psychiatric disorders) | 1 | 0
Executive dysfunction (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 1 | 0
Mood altered (Psychiatric disorders) | 1 | 0
Paranoia (Psychiatric disorders) | 1 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 0
Somnambulism (Psychiatric disorders) | 0 | 1
Stress (Psychiatric disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Paranasal sinus mucosal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 21 | 9
Hypotension (Vascular disorders) | 3 | 0
Haematoma (Vascular disorders) | 3 | 0
Flushing (Vascular disorders) | 2 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 1
Varicose vein (Vascular disorders) | 3 | 0
Essential hypertension (Vascular disorders) | 1 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 1 | 0
Infarction (Vascular disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 1 | 0
Labile hypertension (Vascular disorders) | 0 | 1
Peripheral embolism (Vascular disorders) | 0 | 0
Phlebitis (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1
Visual impairment (Eye disorders) | 8 | 3
Vision blurred (Eye disorders) | 4 | 4
Diplopia (Eye disorders) | 1 | 2
Blindness transient (Eye disorders) | 1 | 1
Cataract (Eye disorders) | 2 | 0
Conjunctival haemorrhage (Eye disorders) | 2 | 0
Eye haemorrhage (Eye disorders) | 1 | 0
Mydriasis (Eye disorders) | 1 | 1
Photopsia (Eye disorders) | 1 | 1
Abnormal sensation in eye (Eye disorders) | 0 | 1
Blepharospasm (Eye disorders) | 0 | 1
Blindness (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Eyelid ptosis (Eye disorders) | 0 | 1
Iridocyclitis (Eye disorders) | 1 | 0
Iritis (Eye disorders) | 1 | 0
Keratitis (Eye disorders) | 1 | 0
Lens disorder (Eye disorders) | 1 | 0
Ocular discomfort (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0
Retinal artery occlusion (Eye disorders) | 0 | 1
Scleritis (Eye disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 2 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Chloasma (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Pemphigus (Skin and subcutaneous tissue disorders) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin depigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Iron deficiency (Metabolism and nutrition disorders) | 1 | 2
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 0
Abnormal weight gain (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperhomocysteinaemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Postprandial hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 5 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 3
Breast pain (Reproductive system and breast disorders) | 1 | 1
Metrorrhagia (Reproductive system and breast disorders) | 2 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 2 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1
Adnexa uteri mass (Reproductive system and breast disorders) | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1
Endometrial disorder (Reproductive system and breast disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Menopausal symptoms (Reproductive system and breast disorders) | 0 | 1
Pelvic discomfort (Reproductive system and breast disorders) | 1 | 0
Polycystic ovaries (Reproductive system and breast disorders) | 1 | 0
Premenstrual dysphoric disorder (Reproductive system and breast disorders) | 1 | 0
Testicular mass (Reproductive system and breast disorders) | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 8 | 4
Tinnitus (Ear and labyrinth disorders) | 6 | 2
Ear pain (Ear and labyrinth disorders) | 2 | 2
Vertigo positional (Ear and labyrinth disorders) | 4 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 2 | 0
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0
Cupulolithiasis (Ear and labyrinth disorders) | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0
Eustachian tube disorder (Ear and labyrinth disorders) | 0 | 1
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 | 0
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 6 | 1
Dysuria (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 1
Stress urinary incontinence (Renal and urinary disorders) | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Haemorrhage urinary tract (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 1
Urine abnormality (Renal and urinary disorders) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Eye naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypothyroidism (Endocrine disorders) | 4 | 1
Thyroid mass (Endocrine disorders) | 1 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 2 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Weight decreased (Investigations) | 2 | 0
Weight increased (Investigations) | 1 | 1
Blood magnesium decreased (Investigations) | 1 | 0
Grip strength decreased (Investigations) | 0 | 1
Heart rate irregular (Investigations) | 1 | 0
Platelet count increased (Investigations) | 1 | 0
Prostatic specific antigen abnormal (Investigations) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 2 | 0
Seasonal allergy (Immune system disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Dental disorder prophylaxis (Surgical and medical procedures) | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 1
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 0
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 1 | 0
Pulmonary arteriovenous fistula (Congenital, familial and genetic disorders) | 1 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of results requires review and approval by REDUCE Publication and Presentation Committee

DOCUMENTS (2):
  • Study Protocol (2016-01-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT00738894/Prot_000.pdf
  • Statistical Analysis Plan (2016-01-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT00738894/SAP_001.pdf